CLINICAL TRIAL: NCT02616406
Title: Assessment of Physical Activity to Determine When Patients Return to Baseline Levels of Activity Following Outpatient Inguinal Hernia Surgery
Brief Title: Objective Measure of Recovery After Outpatient Surgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Karl A. Poterack, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 15-001248
Record Dates: First submitted 2015-11-20; First posted 2015-11-26 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Hernia, Inguinal; Convalescence
Keywords: recovery of function
MeSH Terms: conditions — Hernia, Inguinal; Convalescence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Open repair: Repair group to be monitored with wearable activity monitors pre and post op.
  Interventions: Device: GENEactiv
- Laparoscopic group: Laparoscopic surgical repair group to be monitored with wearable activity monitors pre and post op.
  Interventions: Device: GENEactiv

INTERVENTIONS:
Device: GENEactiv — To wear a monitoring device for a period of time prior to surgery and post surgery

SUMMARY:
This is a study using wearable monitoring devices, patient activity and sleep patterns to monitor pre and post operative following outpatient inguinal hernia surgery to determine when these parameters return to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for outpatient inguinal hernia repair without significant medical comorbidities
* Patients who consent to participating and willing to wear device for designated time period per protocol

Exclusion Criteria:

* History of chronic opioid use
* Inability to speak English
* Inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with inguinal hernia who are to have hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Determine time of return to baseline activity following elective outpatient hernia repair using wearable accelerometers that measure physical movement. | 8 weeks

SECONDARY OUTCOMES:
Determine pain levels on visual analog scale after outpatient hernia repair via telephonic questionnaire. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karl A. Poterack, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials